CLINICAL TRIAL: NCT06268223
Title: The Effect of Home-Based Action Observation Training on Chewing and Swallowing Function in Children With Cerebral Palsy
Brief Title: Home-Based Action Observation Training for Chewing and Swallowing Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Seda Nur Kemer, PT, MSc, PhD Candidate, Academic Lecturer, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/315
Record Dates: First submitted 2024-02-05; First posted 2024-02-20 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Palsy; Chewing Disease; Action Obervation Training
MeSH Terms: conditions — Cerebral Palsy; nigropallidal encephalomalacia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental)
  Interventions: Other: Chewing Exercise Training
- Control Group (Active Comparator)
  Interventions: Other: Chewing Exercise Training

INTERVENTIONS:
Other: Chewing Exercise Training — All groups will implement the Functional Chewing Exercise, consisting of 5 sets per day, 5 days a week, for 12 weeks. Additionally, the study group will participate in an Action Observation Training program, conducted via telerehabilitation, involving 1 set per day, 3 days a week, for 12 weeks, with the guidance of a physiotherapist.

SUMMARY:
The goal of this clinical trial is to investigate the effects of home-based Action Observation Training (AOT) applied together with Functional Chewing Training (FuCT) on chewing and swallowing functions and feeding behavior in children with Cerebral Palsy (CP) who have chewing disorders. The main questions it aims to answer are:

* Is the application of Home-Based AOT together with FuCT effective on chewing function in children with CP?
* Is the application of Home-Based AOT together with FuCT effective on swallowing function in children with CP?
* Is the application of Home-Based AOT together with FuCT effective on feeding behavior in children with CP? Within the scope of the study, children with CP will be divided into two groups as the study group and the control group. All groups will implement FuCT routines, comprising 5 sets per day, 5 days a week, for 12 weeks. Additionally, the study group will be included in an AOT program, conducted via telerehabilitation, for 1 set per day, 3 days a week, for 12 weeks, with the guidance of a physiotherapist. All children with CP will be evaluated at the beginning, after 6 weeks, and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Cerebral Palsy,
* Age between 6 and 18,
* IQ level of 70 or above,
* Having complaints related to chewing function and inability to manage solid food intake
* Feeding orally.

Exclusion Criteria:

* Having a neurodegenerative disease other than Cerebral Palsy
* Having additional chronic illnesses such as systemic diseases, cancer, kidney diseases, gastrointestinal system diseases, etc., that may affect nutritional status,
* Experiencing visual or hearing impairment,
* Using any medication and/or oral device that may affect chewing performance,
* Having received previous chewing and/or swallowing training.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Karaduman Chewing Performance Scale | Up to 12 Weeks
  It is used to determine the chewing performance level. What is the Karaduman chewing performance scale? The Karaduman Chewing Performance Scale is an ordinal scale that is valid, reliable, quick and clinically easy to use to determine the chewing performance level in children with cerebral palsy.
Turkish version of the Mastication Observation and Evaluation Instrument | Up to 12 Weeks
  It is used to evaluate chewing skills.It is a criterion-referenced instrument used to assess individual masticatory skills necessary for efficient intake of solid foods. It contains 8 items that are the basis of masticatory function, including movement of the lips, tongue and jaw, duration of mastication, loss of food or saliva, number of swallows and swallowing coordination. Each item in the scale is scored between 1 and 4, and the lower the total score on the scale, the worse the masticatory function.
Test of Masticating and Swallowing Solids in Children | Up to 12 Weeks
  It is used to quantitatively evaluate the effectiveness of chewing function.This is a norm-referenced, valid and reliable tool for quantitatively assessing the efficiency of masticatory function in children aged 4-18 years. Children are asked to eat a standard biscuit (4.5?×?4.5 cm) as soon as possible, but at a safe speed, and to say "yes" or "ah" when they have finished. The participants will be asked to say the following words and will be video recorded. The videos will be watched by the researcher who will make the evaluations and the duration of eating a standard biscuit, the number of bites, the number of chews and the number of swallows while eating a biscuit will be recorded. The results will be interpreted by comparing with normative data.
Nutrient consistency according toInternational Dysphagia Diet Standardisation Initiative | Up to 12 Weeks
  It is used to determine the highest tolerable food consistency level. The highest level of food consistency that the child can tolerate will be determined by asking the caregiver using the visuals prepared according to this tool.
  The level of difficulty experienced by the child while feeding different food consistencies will be evaluated by asking the caregiver according to VAS. The caregiver will evaluate the level of difficulty experienced in a certain food consistency between 0 and 10. A score of "0" means that my child has no difficulty in consuming this consistency, while "10" means that my child has great difficulty in consuming this consistency.
The Pediatric version of the Eating Assessment Tool | Up to 12 Weeks
  It is used to determine the swallowing related symptom severity. It is a scale developed in collaboration with Hacettepe University and University of California.
  In this study, it was used for symptom-specific assessment and observation in paediatric dysphagia. content validity, internal consistency, test-retest reliability and validity were demonstrated. Ten The total score of the scale consisting of questions varies between 0 and 40 points.
Dysphagia Disorder Survey | Up to 12 Weeks
  It is used to evaluate swallowing function. It is a valid and reliable swallowing disorder assessment tool developed and standardised in child and adult populations diagnosed with intellectual and developmental disabilities. It is based on video-recording and observation of a typical meal in which the child consumes foods appropriate to his/her diet.
Behavioral Pediatrics Feeding Assessment Scale | Up to 12 Weeks
  It is used in the assessment of child feeding behavior. The scale is a 35-question questionnaire that has been culturally adapted and its Turkish validity and reliability have been demonstrated.
  The first 25 questions are about the child's behaviour and the last 10 questions are about the family's feelings or coping strategies. Each item is rated on a 5-point scale (1=never, 5=always).

CONTACTS AND LOCATIONS:
Locations (1):
- Seda Nur Kemer,PT, MSc,PhD Candidate, Lecturer, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No